CLINICAL TRIAL: NCT07071636
Title: A Prospective Study Evaluating Pegylated Interferon Alpha-2b and Nucleos(t)Ide Analogues in Treating Chronic Hepatitis B With or Without Metabolic Dysfunction-Associated Steatotic Liver Disease
Brief Title: Clinical Efficacy of Pegylated Interferon Alpha-2b Combined With Nucleos(t)Ide Analogues in the Treatment of Chronic Hepatitis B Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-242-02
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peg-IFN α-2b combined with NAs (Experimental): received Peg-IFN α-2b combined with NAs Adults aged 18-65 years, regardless of gender; HBsAg-positive for ≥6 months; HBeAg-negative; HBsAg quantification ≤1500 IU/mL; No restriction on HBV DNA quantification; ALT <10×ULN (upper limit of normal, ≤400 IU/L); No prior interferon therapy within the past 1 year; Signed informed consent form obtained;
  Interventions: Drug: Peg-IFN α-2b combined with NAs

INTERVENTIONS:
Drug: Peg-IFN α-2b combined with NAs — Peg-IFN α-2b (1.5 μg/kg/week) combined with NAs

SUMMARY:
Background Chronic hepatitis B (CHB) is a global health issue that affects a large number of patients. There is currently controversy regarding the treatment strategies for CHB patients with metabolic-associated steatoliver disease (MASLD). Therefore, this study aims to conduct a prospective cohort study to compare the therapeutic effects of pegylated interferon α-2b (Peg IFNα-2b) combined with nucleos(t)ide analogues (NAs) in CHB patients with and without MASLD, and to explore the metabolic improvement effects of Peg IFNα-2b treatment in CHB patients with MASLD.

Design This study is a single-center, non-randomized controlled clinical trial. The subjects are CHB patients planned to receive Peg IFNα-2b combined with NAs, who will be naturally divided into two groups based on the presence or absence of MASLD. The study period is from September 15, 2024, to December 31, 2029, with a planned enrollment of 830 patients.

Methods Inclusion Criteria: Adults aged 18 to 65 years, with HBsAg positivity for more than 6 months, HBeAg negativity, HBsAg level ≤1500 IU/ml, ALT <10 ULN (400 IU/L), no interferon treatment in the past year, and signed informed consent.

Grouping Criteria: Patients will be divided into two groups based on the presence or absence of MASLD. MASLD is defined by hepatic steatosis confirmed by imaging or liver biopsy, and the presence of at least one of the following five metabolic factors: BMI ≥23 or waist circumference exceeding the standard, abnormal blood glucose, blood pressure ≥130/85 mmHg, plasma triglycerides ≥1.70 mmol/L, and abnormal plasma high-density lipoprotein cholesterol.

Exclusion Criteria: Pregnant or breastfeeding patients, heavy drinkers, patients with HIV infection, co-infected with other viral hepatitis, patients with liver cirrhosis or hepatocellular carcinoma, severe cardiocerebrovascular or renal diseases, psychiatric abnormalities, abnormal peripheral blood leukocytes or platelet count, interferon allergy, etc.

Withdrawal Criteria: Patients who withdraw informed consent, request to exit, experience severe adverse events, have serious protocol violations, become pregnant, have poor compliance, are lost to follow-up, or whose continued participation in the study is deemed unsafe by the investigator.

Research Endpoints Primary Endpoint: HBsAg clearance rate at 48 weeks of treatment. Secondary Endpoints: Proportion and baseline reduction of HBsAg <1500 IU/ml at the end of treatment, reduction of HBV DNA levels from baseline and proportion below the detection limit, clearance and seroconversion rates of HBeAg in HBeAg-positive patients, and the incidence of cardiovascular disease in MASLD patients at the end of treatment.

Conclusion This study aims to provide evidence for the individualized treatment of CHB patients with MASLD, clarify the impact of MASLD on the treatment response of CHB patients, optimize treatment protocols, increase clinical cure rates, and explore new strategies for improving patients' metabolic functions. Through this study, we hope to provide more precise decision-making support for clinicians, thereby improving patients' quality of life and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria: Adults aged 18-65 years, regardless of gender; HBsAg-positive for ≥6 months; HBeAg-negative; HBsAg quantification ≤1500 IU/mL; No restriction on HBV DNA quantification; ALT <10×ULN (upper limit of normal, ≤400 IU/L); No prior interferon therapy within the past 1 year; Signed informed consent form obtained; Exclusion of comorbid metabolic dysfunction-associated steatotic liver disease (MASLD).

MASLD meets at least one of the following five metabolic criteria:

BMI ≥23 or waist circumference >94 cm (male)/80 cm (female) Fasting plasma glucose ≥5.6 mmol/L or 2-hour postprandial blood glucose ≥7.8 mmol/L or HbA1c ≥5.7% or diagnosis of Type 2 Diabetes Mellitus or undergoing anti-diabetic therapy Blood pressure ≥130/85 mmHg or receiving antihypertensive medication Plasma triglycerides ≥1.70 mmol/L or current lipid-lowering treatment Plasma HDL-C: <1.0 mmol/L (male) or <1.3 mmol/L (female) or active lipid-modifying therapy -

Exclusion Criteria: Patients who are pregnant or breastfeeding. Excessive alcohol consumption: ethanol intake greater than 210g/week for males and greater than 120g/week for females (according to the "Guidelines for the Prevention and Treatment of Metabolic Associated (Non-alcoholic) Fatty Liver Disease (2024 Edition)") Individuals co-infected with HIV. Patients co-infected with HCV virus or other viral hepatitis and other chronic liver diseases.

Patients with liver cirrhosis (compensated or decompensated), liver failure, hepatocellular carcinoma, or any type of malignant tumor.

Patients with serious heart, brain, kidney, and hematopoietic system diseases or oncologic diseases.

Patients with severe psychiatric abnormalities as well as uncontrolled hypertension, diabetes, thyroid dysfunction, etc.

Peripheral blood leukocyte count <3.5×10^9/L and/or platelet count <80×10^9/L. Patients allergic to interferon, as well as those with contraindications to interferon indicated in the package insert.

Patients deemed unsuitable for enrollment by the researcher.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary study endpoint | 48 weeks
  The rate of HBsAg clearance in patients at 48 weeks of treatment.

SECONDARY OUTCOMES:
Secondary study endpoints | 48 weeks
  The proportion of patients with HBsAg <1500 IU/mL and the degree of reduction from baseline at the end of treatment; The degree of reduction in HBV DNA levels from baseline at the end of treatment and the proportion below the detection limit; The proportion of HBeAg-positive patients achieving HBeAg clearance and seroconversion at the end of treatment; The proportion of MASLD patients who develop cardiovascular diseases at the end of treatment.

IPD SHARING:
Plan to Share IPD: No